CLINICAL TRIAL: NCT05455567
Title: OCTA as a New Biomarker in the Pathogenesis of Primary Open Angle Glaucoma
Brief Title: OCTA Study of Choroidal Vasculature in Open Angle Glaucoma Patients
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, professor, Federico II University
Other Study IDs: 0102/22
Record Dates: First submitted 2022-07-07; First posted 2022-07-13 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma Open-Angle Primary
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients with pre perimetric open angle glaucoma
  Interventions: Diagnostic Test: OCTA
- patients with perimetric open angle glaucoma
  Interventions: Diagnostic Test: OCTA
- healthy patients
  Interventions: Diagnostic Test: OCTA

INTERVENTIONS:
Diagnostic Test: OCTA — Choriocapillary vessel density calculated with OCTA

SUMMARY:
The aim of the present study was to examine and measure SFCT and CCVD using respectively EDI-OCT and OCTA in preperimetric and advanced glaucomatous eyes, in order to shed light on the vascular pathogenesis of glaucoma disease.

ELIGIBILITY:
Inclusion Criteria:• age older than 40 years

* diagnosis of glaucoma
* absence of diabetes, heart diseases, hypertension
* absence of drug intake
* absence of vitreoretinal, vascular retinal diseases
* absence of previous ocular surgery and congenital eye diseases.
* absence of errors of refraction
* absence of lens opacities
* absence of low-quality OCT and OCTA images

Exclusion Criteria:

* age younger than 40 years
* presence of diabetes, heart diseases, hypertension
* vitreoretinal and vascular retinal diseases
* previous ocular surgery and congenital eye diseases
* errors of refraction
* lens opacities
* low-quality OCT and OCTA images

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participans were older than 40 years with diagnosis of open angle glaucoma. They did not present any other ophthalmological disease, diabetes, heart diseases and hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
The measurements of choroidal thickness and choriocapillary vessel density in patients with open angle glaucoma. | up to 5 months
  correlation of measurement of choroidal thickness and choriocapillary vessel density in three different patients groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples "Federico II", Naples, Italy

IPD SHARING:
Plan to Share IPD: Yes